CLINICAL TRIAL: NCT03272607
Title: Reducing Post-discharge Adverse Drug Events Amongst the Elderly: a Multi-centre Electronic Deprescribing Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University Health Network, Toronto (Other); The Ottawa Hospital (Other); Foothills Medical Centre (Other); University of Alberta (Other); Kingston Health Sciences Centre (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Emily McDonald, Dr. Emily McDonald, Assistant Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: MedSafer; CIHR Application No. 365795 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Adverse Drug Event
Keywords: Adverse Drug Event; Choosing Wisely Canada; Deprescribing; Elderly; Frailty; High value healthcare; Medication rationalization; Medication stewardship; Polypharmacy
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Frailty

STUDY DESIGN:
Intervention Model Description: The duration of the project will be a total of (approx.) 96 weeks. This is a stepped wedge cluster randomized trial study design (see PDF attachment entitled "MedSafer, Figure 1" - note start date will be August 2017 not July 2016). The intervention component will be administered sequentially to six (6) clusters (by city). A randomly selected single cluster will move from control data collection to intervention data collection every 200 patients or roughly every 12 weeks (96 total weeks), which will be followed by 12 weeks to complete follow up and another 36 to analyze data.
  Please see PDF attachment entitled "MedSafer, Figure 2" which refers to both parts of the study (quality improvement and follow up components). It describes the follow up component of the study (a 30-day telephone follow-up to ascertain adverse drug events- please note the gray-shaded boxes refer to the Quality Improvement Project-Part 1).
Who Masked: Outcomes Assessor
Masking Description: Medical chart abstracts compiled at discharge (including any subsequent visits within 30 days) will be combined with the patient telephone interview into a case summary report which will be reviewed independently by two trained and blinded clinician reviewers who will be made up of pharmacists and physicians from each study site (but who will not adjudicate any patients from their own site).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): All participants in the control arm will receive medication reconciliation at admission and discharge, and identical follow up, but no prioritized deprescribing list will be generated.
- Intervention (Experimental): Participants in the intervention arm will be electronically screened using an electronic software "MedSafer" which will generate output of PIMs that will be brought to the attention of the CTU team via the unit pharmacist as "deprescribing opportunities". (Note that in the case of multiple recommendations, they will be limited and prioritized so as to avoid overwhelming the treating team.) Based on their own expert medical judgement, in collaboration with the patient/caregiver and other relevant clinicians, a decision will be made to deprescribe if appropriate by the patient's in-hospital doctors.
  Interventions: Other: Deprescribing opportunities

INTERVENTIONS:
Other: Deprescribing opportunities — An electronic intervention that identifies potentially inappropriate medications (PIMs) and generates instructions for safe discontinuation, which is presented to the treating physician for their consideration.
  Arms: Intervention

SUMMARY:
Reducing medications and associated side effects in older adults: an electronic hospital-based intervention

DETAILED DESCRIPTION:
Polypharmacy, or the concomitant use of 5 drugs or more, is a serious health concern and affects more than half of Canadians aged 65 years and older. It is the number one identifiable risk factor for adverse drug events (ADEs), which are responsible for 27,000 hospital admissions annually in Canada and up to 20% of return visits to the hospital within 30 days of discharge. Many ADEs are preventable or ameliorable through interventions to reduce inappropriate prescribing.

MedSafer, the intervention software, applies an electronic set of criteria, previously designed and piloted on one thousand (1000) hospitalized patients by a group of Quebec and Ontario internists, geriatricians, palliative care doctors and pharmacists, to identify potentially inappropriate medications (PIMs) in the hospitalized elderly and generate instructions for the patient and physician for safe discontinuation. The current study seeks to partially automate the deprescribing process and to demonstrate the efficacy of this type of intervention on adverse drug events at 30-days post hospital discharge.

At the time of hospitalization, the patient's medications, co-morbidities, and a measure of frailty will be entered into the MedSafer software which will output an individualized and prioritized deprescription plan for the most responsible physician's consideration. Any subsequent medication changes will be transmitted to relevant community physicians. The study will evaluate the impact of stopping PIMs on the occurrence of ADEs within 30 days of discharge, as compared to usual care.

This study will take place on the clinical teaching units (CTUs) at 11 hospitals from seven university hospital centres across Canada. Based on historical data, the investigators estimate a combined 5200 eligible patients per year with nearly 50% taking ten or more medications. Many will have multiple medical co-morbidities such as diabetes, heart disease, and renal insufficiency. A large portion will meet criteria for geriatric syndromes such as frailty and will be at high risk for the development of delirium, falls and functional decline. This population is ideal for a generalizable deprescribing study.

All patients aged 65 or older who meet inclusion/exclusion criteria will be enrolled. A trained research assistant will identify eligible patients and medications will be screened using MedSafer. A deprescribing plan will be generated for the CTU team containing the rationale for suggested medication changes and strategies for safe and successful deprescription. The CTU team will then decide, in conjunction with the patient/proxy and relevant consultants, whether to apply the suggested modifications.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 years and older
* patients who take five or more medications in the community
* patients who are cognitively impaired or otherwise unable to provide consent will still be included as this subpopulation of patients may be at greatest risk of ADEs because of their communication problems.

Exclusion Criteria:

* patients who take four or fewer medications in the community
* patients expected to die within 30 days or be transferred to a palliative care unit/another hospital
* patients without provincial health insurance or who normally live outside that province
* patients previously enrolled
* inability for patient or proxy to speak English or French
* no means of contacting patient or proxy post-discharge

Patients discharged from non-study units will be excluded unless that unit is a transitional care, rehabilitation, or post-acute care unit which bridges the gap between acute medical hospitalization and community services.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6582 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Adverse Drug Events within 30 days post-discharge (ascertained via telephone interviewer and adjudicated via clinician reviewers) | Interview performed 30-35 days post-discharge.
  Post-discharge telephone interview performed by trained personnel using a modification of the Australian two-step adverse reaction and drug event report.
  Two trained and blinded clinician reviewers will independently use the Leape and Bates approach to assess whether an ADE was present (yes/no) and if so what was the nature of the injury resulting from it using a four-point Likert scale (definitely preventable, probably preventable, probably not preventable, and definitely not preventable), and assess the probability that an event was attributable to a specific drug that was newly started, changed or continued during hospitalization. In cases of disagreement, a third trained and blinded clinician will review and determine the final assessment.

SECONDARY OUTCOMES:
Number of potentially inappropriate medications | At hospital discharge and at 30-days post hospital discharge
  The absolute number of potentially inappropriate medications at discharge among patients who were identified as having a potentially inappropriate medication at admission and for who a deprescribing opportunity was generated and presented to the treating team
Mortality within 30-days post discharge | 30-days post hospital discharge
  Death following hospital discharge
Proportion of participants with one or more potentially inappropriate medications deprescribed | At hospital discharge
  Proportion of participants with one or more potentially inappropriate medications deprescribed at discharge between intervention and control
Quality of sleep | 30 days post hospital discharge
  Quality of sleep measured by the PROMIS Sleep Disturbance 4a measured pre- and post-hospitalization compared between intervention and control
Adverse events | 30 days post hospital discharge
  The proportion of patients who had one or more adverse events (falls, hospitalization, death, unplanned encounter with the healthcare system
Falls post hospital discharge | 30 days post hospital
  The proportion of patients with one or more self-reported falls post hospital discharge
Quality of life of participants | At 30-days post hospital discharge
  Quality of life as measured by EQ5D-5L and reported based on reported Canadian time trade-off values (from 0-1 with higher equal to better quality of life)

OTHER OUTCOMES:
Death post hospital discharge | 30-days post hospital discharge
  Proportion of patients who died post-hospital discharge compared between the intervention and control groups
Unplanned visits with the healthcare system | 30-days post hospital discharge
  Proportion of patients with any self-reported unplanned visit with the healthcare system compared between intervention and control (emergency room visits and hospitalizations)
Total number of medications at 30-days | At 30-days post discharge
  Total number of mediations at 30 days (reported as median and interquartile range) compared between intervention and control
Sensitivity analysis for adverse drug events | At 30-days post hospital discharge
  Proportion of participants with 1 or more adverse drug events as defined by 4 or more on the 6-point Leape and Bates Likert scale
Proportion of potentially inappropriate medications that remained stopped | 30-days post hospital discharge
  Proportion of potentially inappropriate medications that remained stopped between intervention and control

CONTACTS AND LOCATIONS:
Overall Officials: Todd C Lee, MD, MPH, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (7):
- Canada (7):
  - Foothills Medical Centre, Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Edmonton, Alberta
  - University of British Columbia, St-Paul's Hospital, Vancouver, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Toronto, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
We will keep a coded, completely anonymized, database that will be made available to other researchers upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Eighteen (18) months following the study completion.

REFERENCES:
- [Derived] McDonald EG, Wu PE, Rashidi B, Wilson MG, Bortolussi-Courval E, Atique A, Battu K, Bonnici A, Elsayed S, Wilson AG, Papillon-Ferland L, Pilote L, Porter S, Murphy J, Ross SB, Shiu J, Tamblyn R, Whitty R, Xu J, Fabreau G, Haddad T, Palepu A, Khan N, McAlister FA, Downar J, Huang AR, MacMillan TE, Cavalcanti RB, Lee TC. The MedSafer Study-Electronic Decision Support for Deprescribing in Hospitalized Older Adults: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2022 Mar 1;182(3):265-273. doi: 10.1001/jamainternmed.2021.7429. PMID 35040926